CLINICAL TRIAL: NCT05283694
Title: A Randomized Open-Label Single Dose Study to Evaluate the Effect of Rate and Volume of Administration on the Bioavailability of Risankizumab Following Subcutaneous (SC) Dosing in Healthy Volunteers
Brief Title: A Study to Evaluate the Bioavailability of Risankizumab Following Subcutaneous Dosing in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M16-324
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Risankizumab Dose A (Experimental): Participants will receive 3 Subcutaneous (SC) injections of risankizumab Dose A administered via prepared syringe at Day 1 and followed for 140 days.
  Interventions: Drug: risankizumab
- Risankizumab Dose B (Experimental): Participants will receive 1 SC injection of risankizumab Dose B administered via syringe pump at Day 1 and followed for 140 days.
  Interventions: Drug: risankizumab
- Risankizumab Dose C (Experimental): Participants will receive 1 SC injection of risankizumab Dose C administered via syringe pump at Day 1 and followed for 140 days.
  Interventions: Drug: risankizumab
- Risankizumab Dose D (Experimental): Participants will receive 1 SC injection of risankizumab Dose D administered via prepared syringe at Day 1 and followed for 140 days.
  Interventions: Drug: risankizumab

INTERVENTIONS:
Drug: risankizumab — Subcutaneous Injection via prepared syringe
  Other Names: ABBV-066; SKYRIZI
  Arms: Risankizumab Dose A; Risankizumab Dose D
Drug: risankizumab — Subcutaneous Injection via syringe pump
  Other Names: ABBV-066; SKYRIZI
  Arms: Risankizumab Dose B; Risankizumab Dose C

SUMMARY:
The objective of this study is to evaluate the bioavailability, safety and tolerability of risankizumab following subcutaneous injections in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Body weight less than 100.00 kg inclusive at Screening and Check-In Day.
* Body Mass Index (BMI) is ≥ 18.0 to ≤ 29.9 kg/m2 after rounded to the tenths decimal, at Screening and upon confinement.

Exclusion Criteria:

* Previous exposure to any anti-IL-12/23 or anti-IL-23 treatment.
* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma), renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Up to 140 Days
  Maximum Observed Plasma Concentration
Time to maximum observed plasma concentration (Tmax) | Up to 140 Days
  Time to maximum observed plasma concentration
Area under the plasma concentration-time curve (AUC) from time 0 to the time of last measurable concentration (AUCt) | Up to 140 Days
  AUC from time 0 to the time of last measurable concentration
AUC from time 0 to infinity (AUCinf) | Up to 140 Days
  AUC from time 0 to infinity
Terminal phase elimination rate constant (β) | Up to 140 Days
  Terminal phase elimination rate constant
Terminal phase elimination half-life (t1/2). | Up to 140 Days
  Terminal phase elimination half-life
Number of Anti-drug antibody (ADA) Titers | Up to 140 Days
  Incidence of anti-drug antibodies
Number of Participants with Adverse Events | Up to 140 Days
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 165737, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No